CLINICAL TRIAL: NCT01899560
Title: Prospective Physiological Study of Lung Elastance in Recruitment and Derecruitment in Early Onset Mechanically Ventilated Acute Respiratory Distress Syndrome (ARDS)Patients
Brief Title: ELASTANCE: Prospective Physiological Study of Lung Elastance in Recruitment and Derecruitment in Early Onset Mechanically Ventilated ARDS Patients
Acronym: ELASTANCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CH-2012-03 2012-A01160-43
Record Dates: First submitted 2013-07-11; First posted 2013-07-15 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Acute respiratory distress syndrome (ARDS); positive end expiratory pressure (PEEP); Staircase recruitment maneuver (SRM); Lung elastance; chest wall elastance
MeSH Terms: conditions — Respiratory Distress Syndrome

ARMS (1):
- Unique arm (Other): Experimental and comparator
  Interventions: Procedure: Measure lung and chest wall elastance with esophageal catheter; Other: non-invasive method for measuring the lung elastance

INTERVENTIONS:
Procedure: Measure lung and chest wall elastance with esophageal catheter — Patients will be in supine position with 30-45° head of bed elevation. The cuff of the endotracheal tube will be transiently overinflated to 60 cmH2O to ensure there will be no air leaks. NMBA (cisatracurium) will be administrated [9]. The fraction of inspired oxygen (FiO2) will be adjusted for continuously monitored oxygen saturation (SpO2) between 90 to 94%. Patients will be ventilated in pressure control with 15 cmH2O of driving pressure.
  A low flow pressure/volume curve from 0 to 40 cmH2O will be performed.
Other: non-invasive method for measuring the lung elastance — by measuring volume recruited during a change of pressure (∆PEEP/∆EELV)

SUMMARY:
The recruitment strategy in Acute respiratory distress syndrome (ARDS) patients mechanically ventilated combines recruitment maneuvers and positive end expiratory pressure (PEEP). Recruitment maneuvers promote alveolar recruitment leading to increased end-expiratory lung volume in order to prevent repetitive opening and closing of unstable lung units and reduce the strain induced by ventilation. In addition, recruitment is effective in improving oxygenation. Variety of recruitment maneuver have been described, the most commonly used is the application of sustained continuous positive airway pressure at 40 cmH2O for 40 seconds. Staircase recruitment maneuver (SRM) is an alternative with good hemodynamic tolerance. Staircase recruitment maneuver (SRM) involves a progressive increase in positive end expiratory pressure (PEEP) (up to 40 cmH2O), in pressure control ventilation, in order to increase end-expiratory lung volume (EELV); then a decreasing PEEP trial is performed. The positive end expiratory pressure (PEEP) to prevent alveolar collapse depends on ratio between lung elastance and chest wall elastance. If chest wall elastance is high, the PEEP to obtain a positive end-expiratory transpulmonary pressure is high. The only way for the time being to know the transpulmonary pressure and the ratio between lung and chest wall elastance is the use of esophageal catheter. A non-invasive method for measuring the lung elastance by measuring volume recruited during a change of pressure (∆PEEP/∆EELV) could be used to avoid the use of esophageal catheter.

ELIGIBILITY:
Inclusion Criteria:

Early onset (less than 24 hours)moderate or severe Acute respiratory distress syndrome (ARDS) according to Berlin Definition

Mechanical ventilation for less than 72 hours

Exclusion Criteria:

Bronchopleural fistula, Emphysema, Pneumothorax, Antecedent of pneumothorax, Increase intracranial pressure, Pulmonary arterial hypertension with right heart failure, Hemodynamic instability with mean arterial pressure < 65 mmHg, Pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2014-11-27 (Actual)

PRIMARY OUTCOMES:
lung and chest wall elastance | 1 Hour
  Measure lung and chest wall elastance with esophageal catheter and compare with the non-invasive method at each level of positive end expiratory pressure (PEEP) during recruitment from 5 to 40 cmH2O and derecruitment from 40 to 5 cmH2O.

SECONDARY OUTCOMES:
Direct volume measurements | 1 Hour
  Determine dynamics of recruitment and derecruitement by direct volume measurements in early onset mechanically ventilated ARDS patients to determine optimal duration and number of breath required for each step during a SRM and a decreasing PEEP trial
the pressure associated with the largest hysteresis on the PV curve | 1 hour
  To set positive end expiratory pressure (PEEP)
The deflection point on the low flow PV curve (ref Hickling AJRCCM 2001), | 1 hour
  To Set positive end expiratory pressure (PEEP)
The minimal PEEP to obtain an positive end-expiratory transpulmonary pressure (ref Talmor NEJM 2009) | 1 Hour
  To set positive end expiratory pressure (PEEP)
- the derecruitment point by SpO2 monitoring during the decreasing positive end expiratory pressure (PEEP)trial (The derecruitment point will be defined as positive end expiratory pressure (PEEP) for which SpO2 decrease) (ref Girgis RC2006). | 1 Hour
  to set positive end expiratory pressure (PEEP)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Intercommunal de Toulon La Seyne sur mer, Toulon, Paca, France